CLINICAL TRIAL: NCT06647810
Title: Relative Bioavailability of Two Different BI 690517 Formulations as Well as the Effect of Multiple Doses of Probenecid on the Single Dose Pharmacokinetics of BI 690517 Following Oral Administration in Healthy Male and Female Subjects (a Randomised, Open-label, Three-way Crossover Trial)
Brief Title: A Study in Healthy People to Test How 2 Different Formulations of BI 690517 Are Taken up in the Body and How Probenecid Influences the Amount of BI 690517 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1378-0025; 2024-513590-45-00 (Registry Identifier: CTIS); U1111-1307-2145 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 690517 formulation 1, then BI 690517 formulation 2, then Probenecid + BI 690517 formulation 2 (Experimental)
  Interventions: Drug: BI 690517 formulation 1; Drug: BI 690517 formulation 2; Drug: Probenecid
- BI 690517 formulation 2, then Probenecid + BI 690517 formulation 2, then BI 690517 formulation 1 (Experimental)
  Interventions: Drug: BI 690517 formulation 1; Drug: BI 690517 formulation 2; Drug: Probenecid
- Probenecid + BI 690517 formulation 2, then BI 690517 formulation 1, then BI 690517 formulation 2 (Experimental)
  Interventions: Drug: BI 690517 formulation 1; Drug: BI 690517 formulation 2; Drug: Probenecid

INTERVENTIONS:
Drug: BI 690517 formulation 1 — BI 690517 formulation 1
  Other Names: Vicadrostat
Drug: BI 690517 formulation 2 — BI 690517 formulation 2
  Other Names: Vicadrostat
Drug: Probenecid — Probenecid
  Other Names: Probenecid Biokanol®

SUMMARY:
This trial aims to test how two different formulations of BI 690517 are taken up by the body and how probenecid influences the amount of BI 690517 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive)
* Signed and dated written informed consent m accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm (beats per minute)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of BI 690517 in plasma over the time interval from 0 to the last quantifiable data point) | Up to day 3.
  For the relative bioavailability of BI 690517.
Cmax (maximum measured concentration of BI 690517 in plasma) | Up to day 3.
  For the relative bioavailability of BI 690517.
AUC0-∞ (area under the concentration-time curve of BI 690517 in plasma over the time interval from 0 extrapolated to infinity) | Up to day 3.
  For the drug interaction of BI 690517 with probenecid.
Cmax (maximum measured concentration of BI 690517 in plasma) | Up to day 3.
  For the drug interaction of BI 690517 with probenecid.

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of BI 690517 in plasma over the time interval from 0 extrapolated to infinity) | Up to day 3.
  For the relative bioavailability of BI 690517.
AUC0-tz (area under the concentration-time curve of BI 690517 in plasma over the time interval from 0 to the last quantifiable data point) | Up to day 3.
  For the drug interaction of BI 690517 with probenecid.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com